CLINICAL TRIAL: NCT03523013
Title: The Outcome of CPAP Titration Under Sleep Endoscopy: A Randomized Controlled Crossover Trial
Brief Title: The Outcome of CPAP Titration Under Sleep Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 201701422A3
Record Dates: First submitted 2018-03-26; First posted 2018-05-14 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2018-02

CONDITIONS: Obstructive Sleep Apnea; CPAP; DISE
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPAP pressure (determied by DISE) (Experimental)
  Interventions: Device: CPAP
- CPAP pressure (determined by physician) (Active Comparator)
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP — CPAP treatment with different pressure for OSA patients

SUMMARY:
The outcome of CPAP titration under sleep endoscopy: A randomized controlled crossover trial

DETAILED DESCRIPTION:
This is the study entitled "The outcome of CPAP titration under sleep endoscopy: A randomized controlled crossover trial". CPAP is first line golden standard treatment for Obstructive sleep apnea (OSA). However, the overall CPAP compliance is about 50%. One of the reasons responsible for the poor compliance is the inadequate pressure setting initially. Therefore, it is crucial for us to find out the adequate pressure as soon as possible. Sleep endoscopy is the way to evaluate upper airway obstruction of OSA patients. Meanwhile, the investigators used CPAP to titrate the adequate pressure to keep upper airway open under sleep endoscopy guidance. While the investigators find out this adequate pressure, the investigators set this pressure into CPAP program, which OSA patient will use for 1 month. To compare the different effect of CPAP under either auto-CPAP titration pressure or sleep endoscopy guidance pressure, those OSA patients will use auto-titration CPAP for 1 month as well. Another highlight of this study is the sedative agent-dexmedetomidine. Dexmedetomidine is a α2 antogonist, which cause patients sedative but less respiratory drive suppression. The mechanism of dexmedetomidine is more physiological for nature sleep.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe OSA
* ESS >10

Exclusion Criteria:

* ASA > 3
* allergy to Dexmedetomidine
* second or third degree AVB
* severe heart failure Fc class IV
* asthma acute attack

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
complaince of CPAP use | the change of complaince between baseline, 1 month and 2 months
  CPAP complaince was defined as the use of CPAP is more than 4 hours per day and 5 days per week

SECONDARY OUTCOMES:
sleepiness score | the change of ESS between baseline, 1 month and 2 months
  ESS

OTHER OUTCOMES:
sleep quality | the change of PSQ between baseline, 1 month and 2 months
  PSQ

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Thoracic Medicine, Chang Gung Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang TY, Huang YC, Lin TY, Ni YL, Lo YL. Outcome of CPAP Titration for Moderate-to-Severe OSA Under Drug-Induced Sleep Endoscopy: A Randomized Controlled Crossover Trial. Front Neurol. 2022 Jun 13;13:882465. doi: 10.3389/fneur.2022.882465. eCollection 2022. PMID 35769360